CLINICAL TRIAL: NCT00583947
Title: A Cumulative Dose Safety and Tolerability Crossover Study of Arformoterol Tartrate Inhalation Solution and Levalbuterol Hydrochloride Inhalation Solution in Pediatric Subjects (Aged 2 to 11 Years of Age) With Asthma
Brief Title: A Safety and Tolerability Study of Arformoterol Tartrate Inhalation Solution in Pediatric Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 091-029
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
Keywords: Asthma; Respiratory Tract Diseases
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases | interventions — Formoterol Fumarate; Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARF/LEV (Other): Cross-over phase: one day active treatment with arformoterol 7.5 microgram per nebulization followed by a 7 day washout. Then a one day active treatment with levalbuterol 0.63 milligram per nebulization.
  Open-label phase: Following another 7 day washout, one day treatment with arformoterol 15 micrograms per nebulization.
  Interventions: Drug: arformoterol; Drug: levalbuterol
- LEV/ARF (Other): Cross-over phase: one day active treatment with levalbuterol 0.63 milligram per nebulization followed by a 7 day washout. Then a one day active treatment with arformoterol 7.5 micrograms per nebulization.
  Open-label phase: Following another 7 day washout, one day treatment with arformoterol 15 micrograms per nebulization.
  Interventions: Drug: arformoterol; Drug: levalbuterol

INTERVENTIONS:
Drug: arformoterol — Arformoterol is given at a 7.5 ug per dosing during the cross-over phase and 15 ug per dosing during the open-label phase. Each treatment consists of one nebulization every 30 minutes over a 60 minute treatment interval (totaling 3 cumulative dosings at 0,30 and 60 minutes).
  Other Names: Brovana
Drug: levalbuterol — Levalbuterol is given at a 0.63 mg per dosing during the cross-over phase. Each treatment consists of one nebulization every 30 minutes over a 60 minute treatment interval (totaling 3 cumulative dosings at 0,30 and 60 minutes).
  Other Names: Xopenex

SUMMARY:
To determine the safety and tolerability of Arformoterol Tartrate in children with asthma

DETAILED DESCRIPTION:
A randomized, double-blind two-way crossover study of three cumulative doses of arformoterol (7.5 ug per nebulization) and levalbuterol (0.63 mg per nebulization) given over a one hour period, followed by a single open-label treatment day with three cumulative doses of arformoterol 15 ug in subjects 2-11 years of age with asthma. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Between Age 2 and 11, inclusive, at the time of consent
* Weight equal to or greater than 15 Kg
* History of physician-diagnosed asthma of at least 2 years duration for children age 6 and older, and at least 1 year duration for children 5 and younger.

Exclusion Criteria:

* Female subject who is pregnant or lactating.
* Subject who has a history of hospitalization for asthma within one year, or who is scheduled for in-patient hospitalization, including elective surgery during the course of the trial.
* Subject with any history of life-threatening asthma defined as a history of asthma episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* Subject with a history of cancer.
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders.
* Subject with a history of cigarette smoking or use of any tobacco products.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pulmonary Medical Director, Study Chair — Unicorn Pharma Consulting
Locations (13):
- United States (13):
  - Beverly Hills, California
  - Orange, California
  - Savannah, Georgia
  - Normal, Illinois
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Upland, Pennsylvania
  - Orangeburg, South Carolina
  - Spartanburg, South Carolina
  - Dallas, Texas
  - Burke, Virginia
  - Richmond, Virginia

REFERENCES:
- [Result] Hinkle J, Hinson J, Kerwin E, Goodwin E, Sciarappa K, Curry L, Hanrahan JP. A cumulative dose, safety and tolerability study of arformoterol in pediatric subjects with stable asthma. Pediatr Pulmonol. 2011 Aug;46(8):761-9. doi: 10.1002/ppul.21446. Epub 2011 May 16. PMID 21584948

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 86 subjects were screened: 23 subjects aged 2-5 years and 63 subjects aged 6-11 years.
Groups:
- ARF/LEV: Cross-over period: one day active treatment with arformoterol 7.5 microgram per nebulization followed by a 7 day washout. Then a one day active treatment with levalbuterol 0.63 milligram per nebulization.
  Open-label period: Following another 7 day washout, one day treatment with arformoterol 15 micrograms per nebulization.
- LEV/ARF: Cross-over period: one day active treatment with levalbuterol 0.63 milligram per nebulization followed by a 7 day washout. Then a one day active treatment with arformoterol 7.5 micrograms per nebulization.
  Open-label period: Following another 7 day washout, one day treatment with arformoterol 15 micrograms per nebulization.
Period: Cross-over Period
Arm/Group | ARF/LEV | LEV/ARF
Started | 27 (Participants were stratified by age group at randomization: ages 2-5 yrs and 6-11 years) | 26 (Participants were stratified by age group at randomization: ages 2-5 yrs and 6-11 years)
Completed | 22 | 24
Not Completed | 5 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Did not meet-no longer met entry criteri | 0 | 1
Not completed — Other | 1 | 1
Period: Washout
Arm/Group | ARF/LEV | LEV/ARF
Started | 22 | 24
Completed | 22 | 24
Not Completed | 0 | 0
Period: Open Label Period
Arm/Group | ARF/LEV | LEV/ARF
Started | 22 (3 subjects were dosed with arformoterol 7.5 microgram in error) | 24 (3 subjects were dosed with arformoterol 7.5 microgram in error)
Completed | 22 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARF/LEV: Cross-over: Participants treated with arformoterol 7.5 microgram per nebulization; 7 day washout; levalbuterol 0.63 milligram per nebulization.
  Open label: 7 day washout; arformoterol 15 microgram per nebulization.
- LEV/ARF: Cross-over: Participants treated with levalbuterol 0.63 milligram per nebulization; 7 day washout; arformoterol 7.5 microgram per nebulization.
  Open label: 7 day washout; arformoterol 15 microgram per nebulization.
- Total: Total of all reporting groups
Arm/Group | ARF/LEV | LEV/ARF | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 26 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years]
  Age 2-5 years | 4.4 (0.79) | 4.4 (0.79) | 4.4 (0.76)
  Age 6-11 years | 9.0 (1.26) | 8.5 (1.43) | 8.8 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 19 | 12 | 31
  Black/African American | 6 | 14 | 20
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 53
Height [Mean (Standard Deviation); unit: centimeters] | 131.62 (15.244) | 130.42 (15.377) | 131.03 (15.174)
Weight [Mean (Standard Deviation); unit: kilograms] | 31.57 (12.106) | 32.68 (12.802) | 32.12 (12.345)

OUTCOME MEASURES:

1. Primary Outcome: Mean Heart Rate
Description: Heart rate measured at various timepoints: predose and timepoints after each of the three dosings. Each treatment consists of one nebulization every 30 minutes over a 60 minute treatment interval (totaling 3 cumulative dosings at 0,30 and 60 minutes).
Time Frame: predose, various timeframes up to 5 hours post last dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Levalbuterol 0.63 mg: Values represent participant experience when treated with levalbuterol during the cross-over portion of the study
- Arformoterol 7.5 Mcg: Values represent the experience of participants when treated with arformoterol 7.5 mcg during the cross-over portion of the study
- Arformoterol 15 Mcg: Values represent the experience of participants when treated with arformoterol 15 mcg during the open-label portion of the study
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
beats per minute
  Predose (n=51,52,40) | 87.6 (12.56) | 84.7 (14.11) | 87.0 (17.47)
  15 min post dose 1 (n=51,52,40) | 89.3 (15.57) | 85.2 (15.19) | 89.4 (16.88)
  30 min post dose 1 (n=51,52,40) | 90.9 (14.47) | 86.6 (14.63) | 89.5 (15.59)
  60 min post dose 1 (n=51,51,40) | 96.4 (12.33) | 89.0 (13.67) | 93.5 (16.41)
  15 min post dose 2 (n=50,51,40) | 95.4 (12.94) | 87.5 (14.88) | 92.5 (18.60)
  30 min post dose 2 (n=47,50,40) | 97.1 (13.28) | 88.9 (13.33) | 93.3 (16.72)
  60 min post dose 2 (n=46,50,37) | 100.4 (16.60) | 89.3 (13.97) | 96.1 (12.80)
  30 min post last dose (n=49,52,40) | 99.2 (17.38) | 90.3 (14.24) | 96.1 (13.92)
  60 min post last dose (n=49,52,40) | 96.0 (16.45) | 93.3 (13.06) | 97.1 (14.95)
  1.5 hours post last dose (n=48,52,40) | 96.2 (17.29) | 91.8 (11.75) | 95.3 (16.42)
  2 hours post last dose (n=50,52,40) | 93.0 (16.23) | 91.2 (11.77) | 95.9 (14.57)
  2.5 hours post last dose (n=49,52,40) | 94.1 (16.22) | 90.2 (14.61) | 94.8 (15.66)
  3 hours post last dose (n=50,52,40) | 94.1 (14.84) | 90.6 (13.57) | 93.4 (16.04)
  3.5 hours post last dose (n=50,52,40) | 93.3 (14.65) | 89.8 (13.20) | 95.0 (15.16)
  4 hours post last dose (n=50,52,40) | 94.0 (12.68) | 89.3 (11.76) | 94.5 (14.94)
  4.5 hours post last dose (n=50,52,40) | 93.3 (13.71) | 89.6 (12.50) | 93.9 (16.49)
  5 hours post last dose (n=50,51,40) | 92.4 (15.36) | 89.8 (14.16) | 92.9 (14.51)

2. Secondary Outcome: Mean Forced Expiratory Volume in One Second(FEV1)
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer.
Time Frame: predose, various postdose times
Population: Intent to treat population. Pulmonary function testing was only performed on subjects six years of age or older; there were no subjects five or younger who performed spirometry. Subject data for those who were misdosed with ARF 7.5mcg rather than ARF 15mcg in the open-label portion were excluded from these analyses.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 37 | 38 | 27
liters
  predose (n=37,38,27) | 1.554 (0.374) | 1.552 (0.377) | 1.486 (0.294)
  10 minutes post dose 1 (n=37,38,27) | 1.714 (0.411) | 1.668 (0.403) | 1.620 (0.315)
  25 minutes post dose 1 (n=37,37,27) | 1.712 (0.425) | 1.695 (0.409) | 1.644 (0.334)
  10 minutes post dose 2 (n=36,38,27) | 1.741 (0.430) | 1.721 (0.420) | 1.661 (0.332)
  25 minutes post dose 2 (n=36,38,27) | 1.735 (0.438) | 1.714 (0.423) | 1.669 (0.331)
  10 minutes post dose 3 (n=34,38,27) | 1.775 (0.402) | 1.731 (0.419) | 1.689 (0.340)
  25 minutes post dose 3 (n=35,38,26) | 1.782 (0.415) | 1.740 (0.419) | 1.700 (0.345)
  2 hours post dose 1 (n=36,37,27) | 1.784 (0.397) | 1.754 (0.408) | 1.704 (0.337)
  4 hours post dose 1 (n=36,38,27) | 1.732 (0.401) | 1.722 (0.423) | 1.684 (0.344)
  6 hours post dose 1 (n=36,38,27) | 1.667 (0.400) | 1.725 (0.426) | 1.660 (0.356)

3. Primary Outcome: Change From Predose in Mean Heart Rate
Description: Heart rate measured at various timepoints minus the heart rate at predose.
Time Frame: predose, various timeframes up to 5 hours post last dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
beats per minute
  15 min post dose 1 (n=51,52,40) | 1.6 (10.27) | 0.5 (9.40) | 2.3 (10.33)
  30 min post dose 1 (n=51,52,40) | 3.2 (11.91) | 2.0 (11.06) | 2.5 (11.14)
  60 min post dose 1 (n=51,51,40) | 8.7 (10.70) | 4.4 (11.85) | 6.5 (12.62)
  15 min post dose 2 (n=50,51,40) | 7.8 (10.72) | 2.8 (11.48) | 5.5 (12.89)
  30 min post dose 2 (n=47,50,40) | 10.0 (10.67) | 4.5 (10.46) | 6.3 (12.90)
  60 min post dose 2 (n=46,50,37) | 13.2 (13.81) | 4.7 (10.50) | 9.5 (12.89)
  30 min post last dose (n=49,52,40) | 11.9 (14.11) | 5.6 (11.44) | 9.0 (13.34)
  60 min post last dose (n=49,52,40) | 8.7 (13.97) | 8.6 (14.06) | 10.0 (14.81)
  1.5 hours post last dose (n=48,52,40) | 8.9 (11.73) | 7.1 (12.65) | 8.3 (15.95)
  2 hours post last dose (n=50,52,40) | 5.6 (12.13) | 6.6 (10.77) | 8.9 (12.69)
  2.5 hours post last dose (n=49,52,40) | 6.8 (11.20) | 5.5 (14.33) | 7.8 (13.36)
  3 hours post last dose (n=50,52,40) | 6.7 (10.94) | 5.9 (12.74) | 6.4 (13.31)
  3.5 hours post last dose (n=50,52,40) | 5.9 (11.89) | 5.1 (11.63) | 7.9 (12.11)
  4 hours post last dose (n=50,52,40) | 6.6 (10.30) | 4.6 (13.51) | 7.4 (11.62)
  4.5 hours post last dose (n=50,52,40) | 5.9 (10.86) | 4.9 (12.00) | 6.9 (12.70)
  5 hours post last dose (n=50,51,40) | 5.0 (12.03) | 5.3 (12.41) | 5.8 (12.55)

4. Primary Outcome: Mean Systolic Blood Pressure
Description: Systolic blood pressure measured at various timepoints: predose and timepoints after each of the three dosings. Each treatment consists of one nebulization every 30 minutes over a 60 minute treatment interval (totaling 3 cumulative dosings at 0,30 and 60 minutes).
Time Frame: predose, various timeframes up to 5 hours post last dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
mmHg
  Predose (n=51,52,40) | 102.1 (10.80) | 101.5 (9.86) | 100.6 (10.36)
  15 min post dose 1 (n=51,52,40) | 102.9 (10.90) | 101.2 (11.07) | 102.6 (11.42)
  30 min post dose 1 (n=51,52,40) | 104.6 (12.08) | 102.5 (10.20) | 100.3 (9.78)
  60 min post dose 1 (n=51,51,40) | 105.8 (9.31) | 102.7 (9.82) | 103.2 (10.82)
  15 min post dose 2 (n=50,51,40) | 105.0 (11.20) | 101.7 (9.42) | 102.1 (12.20)
  30 min post dose 2 (n=47,50,40) | 106.4 (10.32) | 102.8 (9.26) | 101.9 (9.81)
  60 min post dose 2 (n=46,50,37) | 107.2 (12.05) | 101.9 (11.18) | 102.9 (9.95)
  30 min post last dose (n=49,52,40) | 105.0 (12.22) | 101.2 (11.72) | 101.6 (12.60)
  60 min post last dose (n=49,52,40) | 106.1 (10.32) | 103.0 (11.87) | 104.9 (11.03)
  1.5 hours post last dose (n=48,52,40) | 104.8 (11.43) | 101.9 (11.67) | 103.0 (10.35)
  2 hours post last dose (n=50,52,40) | 104.6 (11.40) | 103.4 (10.81) | 101.8 (10.87)
  2.5 hours post last dose (n=49,52,40) | 103.0 (12.41) | 101.5 (10.58) | 101.3 (10.10)
  3 hours post last dose (n=50,52,40) | 106.1 (12.28) | 102.1 (10.84) | 101.9 (11.57)
  3.5 hours post last dose (n=50,52,40) | 103.4 (10.00) | 103.2 (11.38) | 101.4 (9.41)
  4 hours post last dose (n=50,52,40) | 103.6 (11.26) | 102.1 (10.14) | 100.5 (10.48)
  4.5 hours post last dose (n=50,52,40) | 104.5 (10.50) | 103.2 (10.96) | 101.5 (9.25)
  5 hours post last dose (n=50,52,40) | 106.7 (9.94) | 104.1 (10.46) | 102.1 (9.49)

5. Primary Outcome: Change From Predose in Mean Systolic Blood Pressure
Description: Mean systolic blood pressure measured at various timepoints minus the mean systolic blood pressure at predose
Time Frame: predose, various timeframes up to 5 hours post last dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
mmHg
  15 min post dose 1 (n=51,52,40) | 0.8 (10.58) | -0.4 (9.57) | 2.0 (8.06)
  30 min post dose 1 (n=51,52,40) | 2.6 (10.14) | 0.9 (6.97) | -0.3 (7.68)
  60 min post dose 1 (n=51,51,40) | 3.7 (8.60) | 1.1 (9.54) | 2.6 (7.97)
  15 min post dose 2 (n=50,51,40) | 2.6 (8.94) | -0.3 (9.28) | 1.6 (9.07)
  30 min post dose 2 (n=47,50,40) | 3.3 (8.59) | 0.8 (9.01) | 1.4 (7.19)
  60 min post dose 2 (n=46,50,37) | 4.0 (7.89) | -0.3 (8.98) | 1.8 (8.87)
  30 min post last dose (n=49,52,40) | 2.4 (10.72) | -0.4 (9.37) | 1.1 (11.25)
  60 min post last dose (n=49,52,40) | 3.5 (10.92) | 1.5 (11.17) | 4.4 (8.43)
  1.5 hours post last dose (n=48,52,40) | 1.8 (9.70) | 0.3 (10.22) | 2.4 (8.06)
  2 hours post last dose (n=50,52,40) | 2.3 (10.31) | 1.8 (10.18) | 1.3 (9.44)
  2.5 hours post last dose (n=49,52,40) | 0.4 (10.12) | -0.0 (8.80) | 0.7 (7.77)
  3 hours post last dose (n=50,52,40) | 3.9 (10.58) | 0.6 (8.83) | 1.3 (7.28)
  3.5 hours post last dose (n=50,52,40) | 1.2 (8.87) | 1.7 (10.18) | 0.9 (7.06)
  4 hours post last dose (n=50,52,40) | 1.3 (11.08) | 0.6 (10.17) | -0.0 (8.36)
  4.5 hours post last dose (n=50,52,40) | 2.2 (10.37) | 1.7 (9.61) | 0.9 (8.26)
  5 hours post last dose (n=50,52,40) | 4.5 (10.79) | 2.5 (8.90) | 1.6 (9.62)

6. Primary Outcome: Mean Diastolic Blood Pressure
Description: Diastolic blood pressure measured at various timepoints: predose and timepoints after each of the three dosings. Each treatment consists of one nebulization every 30 minutes over a 60 minute treatment interval (totaling 3 cumulative dosings at 0,30 and 60 minutes).
Time Frame: predose, various timeframes up to 5 hours post last dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
mmHg
  Predose (n=51,52,40) | 62.5 (8.19) | 63.2 (6.82) | 63.6 (9.77)
  15 min post dose 1 (n=51,52,40) | 61.4 (9.32) | 62.0 (7.29) | 62.5 (8.52)
  30 min post dose 1 (n=51,52,40) | 60.8 (8.34) | 62.5 (7.61) | 61.6 (7.56)
  60 min post dose 1 (n=51,51,40) | 63.4 (7.72) | 62.5 (7.47) | 62.3 (9.38)
  15 min post dose 2 (n=50,51,40) | 61.7 (8.76) | 63.3 (6.75) | 60.8 (8.81)
  30 min post dose 2 (n=47,50,40) | 63.1 (7.35) | 62.2 (7.61) | 61.7 (8.86)
  60 min post dose 2 (n=46,50,37) | 62.8 (8.07) | 62.0 (8.15) | 62.3 (7.99)
  30 min post last dose (n=49,52,40) | 63.4 (7.27) | 62.0 (8.83) | 61.6 (7.91)
  60 min post last dose (n=49,52,40) | 63.5 (8.88) | 62.1 (8.60) | 62.5 (8.09)
  1.5 hours post last dose (n=48,52,40) | 63.1 (9.09) | 62.3 (7.90) | 62.5 (9.03)
  2 hours post last dose (n=50,52,40) | 63.8 (10.79) | 62.3 (6.87) | 62.1 (9.62)
  2.5 hours post last dose (n=49,52,40) | 60.7 (10.41) | 59.7 (7.97) | 62.3 (8.71)
  3 hours post last dose (n=50,52,40) | 63.2 (8.85) | 61.4 (7.51) | 62.5 (9.77)
  3.5 hours post last dose (n=50,52,40) | 62.0 (9.80) | 60.5 (6.54) | 62.6 (7.59)
  4 hours post last dose (n=50,52,40) | 62.9 (10.15) | 63.1 (7.32) | 59.9 (8.65)
  4.5 hours post last dose (n=50,52,40) | 62.6 (9.12) | 62.2 (7.84) | 61.9 (8.38)
  5 hours post last dose (n=50,52,40) | 62.3 (8.75) | 63.0 (7.40) | 60.0 (8.59)

7. Primary Outcome: Change From Predose in Mean Diastolic Blood Pressure
Description: Mean diastolic blood pressure measured at various timepoints minus the predose diastolic blood pressure
Time Frame: predose, various timeframes up to 5 hours post last dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
mmHg
  15 min post dose 1 (n=51,52,40) | -1.1 (8.60) | -1.1 (7.26) | -1.0 (10.23)
  30 min post dose 1 (n=51,52,40) | -1.7 (7.69) | -0.6 (7.84) | -1.9 (7.27)
  60 min post dose 1 (n=51,51,40) | 0.8 (7.89) | -0.7 (7.71) | -1.3 (9.43)
  15 min post dose 2 (n=50,51,40) | -1.1 (8.10) | 0.1 (6.85) | -2.8 (9.65)
  30 min post dose 2 (n=47,50,40) | 0.8 (7.82) | -1.1 (7.59) | -1.9 (9.59)
  60 min post dose 2 (n=46,50,37) | 0.0 (7.08) | -1.3 (6.98) | -1.8 (6.91)
  30 min post last dose (n=49,52,40) | 0.8 (7.12) | -1.2 (7.34) | -1.9 (9.35)
  60 min post last dose (n=49,52,40) | 0.8 (8.84) | -1.1 (8.48) | -1.1 (8.31)
  1.5 hours post last dose (n=48,52,40) | 0.1 (8.00) | -0.9 (7.23) | -1.1 (9.38)
  2 hours post last dose (n=50,52,40) | 1.4 (10.16) | -0.9 (7.70) | -1.5 (9.39)
  2.5 hours post last dose (n=49,52,40) | -1.9 (8.66) | -3.5 (7.36) | -1.3 (9.56)
  3 hours post last dose (n=50,52,40) | 0.8 (8.45) | -1.8 (8.31) | -1.1 (10.49)
  3.5 hours post last dose (n=50,52,40) | -0.4 (8.36) | -2.6 (6.66) | -1.0 (8.87)
  4 hours post last dose (n=50,52,40) | 0.5 (10.38) | -0.0 (7.63) | -3.7 (10.29)
  4.5 hours post last dose (n=50,52,40) | 0.2 (8.86) | -1.0 (7.64) | -1.7 (10.42)
  5 hours post last dose (n=50,52,40) | -0.1 (8.84) | -0.1 (8.06) | -3.6 (10.25)

8. Primary Outcome: Mean Serum Potassium Levels
Time Frame: Predose, 2 hours and 6 hours postdose 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 39
mEq/L
  Predose (n=51,52,39) | 4.25 (0.376) | 4.27 (0.386) | 4.31 (0.325)
  2 hours post dose 1 (n=48,47,38) | 3.67 (0.423) | 3.83 (0.391) | 3.71 (0.410)
  6 hours post dose 1 (n=48,49,38) | 3.99 (0.334) | 3.95 (0.325) | 3.87 (0.435)

9. Primary Outcome: Change From Predose in Mean Serum Potassium
Description: Change in mean serum potassium at the specified timepoint minus the predose value.
Time Frame: predose, 2 and 6 hours post dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 39
mEq/L
  2 hours post dose 1 (n=48,47,38) | -0.58 (0.457) | -0.42 (0.407) | -0.62 (0.401)
  6 hours post dose 1 (n=48,49,38) | -0.23 (0.307) | -0.31 (0.450) | -0.39 (0.424)

10. Primary Outcome: Mean Serum Glucose Values
Time Frame: Predose, 2 and 6 hours post dose 1
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
mg/dl
  Predose (n=51,52,40) | 86.4 (15.59) | 87.5 (15.43) | 87.6 (17.41)
  2 hours post dose 1 (n=48,47,39) | 114.5 (30.42) | 108.6 (27.51) | 120.6 (32.52)
  6 hours post dose 1 (n=49,48,38) | 107.6 (18.43) | 99.0 (15.78) | 106.3 (15.64)

11. Primary Outcome: Change From Predose in Mean Serum Glucose
Description: Change in mean serum glucose at the specified timepoint minus the predose value.
Time Frame: predose, 2 and 6 hours post dose
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 40
mg/dl
  2 hours post dose 1 (n=48,47,39) | 27.1 (34.74) | 22.4 (32.66) | 32.9 (35.21)
  6 hours post dose 1 (n=49,48,38) | 20.3 (22.49) | 12.1 (20.59) | 18.6 (23.11)

12. Secondary Outcome: Change From Predose of Mean Forced Expiratory Volume in One Second (FEV1)
Description: Forced Expiratory Volume in one second (FEV1) is the volume of air forcibly exhaled in one second as measured by a spirometer. Change in FEV1 was calculated as postdose value minus the predose value at each visit.
Time Frame: predose, various postdose timepoints
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 37 | 38 | 27
liters
  10 minutes post dose 1 (n=37,38,27) | 0.160 (0.102) | 0.117 (0.112) | 0.133 (0.105)
  25 minutes post dose 1 (n=37,37,27) | 0.159 (0.139) | 0.142 (0.151) | 0.158 (0.125)
  10 minutes post dose 2 (n=36,38,27) | 0.199 (0.130) | 0.169 (0.154) | 0.175 (0.106)
  25 minutes post dose 2 (n=36,38,27) | 0.194 (0.153) | 0.162 (0.166) | 0.183 (0.137)
  10 minutes post dose 3 (n=34,38,27) | 0.226 (0.144) | 0.179 (0.160) | 0.203 (0.148)
  25 minutes post dose 3 (n=35,38,26) | 0.226 (0.154) | 0.188 (0.150) | 0.205 (0.152)
  2 hours post dose 1 (n=36,37,27) | 0.216 (0.139) | 0.194 (0.146) | 0.218 (0.149)
  4 hours post dose 1 (n=36,38,27) | 0.163 (0.150) | 0.170 (0.175) | 0.198 (0.150)
  6 hours post dose 1 (n=36,38,27) | 0.098 (0.128) | 0.173 (0.165) | 0.174 (0.166)

13. Secondary Outcome: Mean Peak Expiratory Flow Rate (PEFR)
Description: PEFR is the fastest rate at which air can move through the airways during a forced expiration starting with fully inflated lungs as measured by peak flow meters.
Time Frame: predose, various postdose times
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 37 | 38 | 27
liters/second
  predose (n=37,38,27) | 3.604 (0.949) | 3.546 (0.928) | 3.565 (0.675)
  10 minutes post dose 1 (n=37,38,27) | 3.926 (0.900) | 3.788 (0.950) | 3.824 (0.613)
  25 minutes post dose 1 (n=37,37,27) | 4.003 (0.893) | 3.877 (0.950) | 3.844 (0.698)
  10 minutes post dose 2 (n=36,38,27) | 4.053 (1.007) | 3.890 (0.998) | 3.925 (0.679)
  25 minutes post dose 2 (n=36,38,27) | 4.047 (0.982) | 3.964 (0.912) | 3.989 (0.652)
  10 minutes post dose 3 (n=34,38,27) | 4.156 (0.960) | 4.003 (0.993) | 4.077 (0.711)
  25 minutes post dose 3 (n=35,38,26) | 4.176 (0.966) | 4.007 (0.899) | 4.017 (0.693)
  2 hours post dose 1 (n=36,37,27) | 4.221 (0.961) | 4.178 (1.013) | 4.066 (0.668)
  4 hours post dose 1 (n=36,38,27) | 4.155 (0.984) | 4.029 (1.061) | 4.039 (0.663)
  6 hours post dose 1 (n=36,38,27) | 3.970 (0.938) | 4.058 (1.075) | 4.016 (0.628)

14. Secondary Outcome: Change From Predose in Mean Peak Expiratory Flow Rate (PEFR)
Description: PEFR is the fastest rate at which air can move through the airways during a forced expiration starting with fully inflated lungs as measured by peak flow meters. Change in PEFR was calculated as postdose value minus the predose value at each visit.
Time Frame: predose, various postdose times
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 37 | 38 | 27
liters/second
  10 minutes post dose 1 (n=37,38,27) | 0.322 (0.305) | 0.242 (0.298) | 0.259 (0.396)
  25 minutes post dose 1 (n=37,37,27) | 0.399 (0.367) | 0.320 (0.392) | 0.279 (0.442)
  10 minutes post dose 2 (n=36,38,27) | 0.458 (0.363) | 0.344 (0.369) | 0.360 (0.406)
  25 minutes post dose 2 (n=36,38,27) | 0.452 (0.329) | 0.419 (0.363) | 0.424 (0.383)
  10 minutes post dose 3 (n=34,38,27) | 0.524 (0.343) | 0.457 (0.439) | 0.513 (0.466)
  25 minutes post dose 3 (n=35,38,26) | 0.539 (0.375) | 0.462 (0.429) | 0.449 (0.497)
  2 hours post dose 1 (n=36,37,27) | 0.575 (0.385) | 0.596 (0.596) | 0.501 (0.408)
  4 hours post dose 1 (n=36,38,27) | 0.509 (0.345) | 0.484 (0.440) | 0.474 (0.449)
  6 hours post dose 1 (n=36,38,27) | 0.324 (0.337) | 0.513 (0.720) | 0.451 (0.462)

15. Secondary Outcome: Plasma Concentration of (R,R) Formoterol
Description: If the mean plasma concentration was 'below the limit of quantification' (BLQ) which was set as <=0.5 picograms/milliliter, the value is displayed as a zero.
Time Frame: predose, various postdose times
Population: PK population consisted of subjects who were in the intent-to-treat population and had any plasma concentration data available.
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Number analyzed (Participants) | 51 | 52 | 39
picogram/milliliter
  predose (n=51,52,39) | 0.646 (3.4172) | 0 (0.5159) | 0.737 (2.7612)
  25 minutes post dose 1 (n=50,46,36) | 2.402 (15.1253) | 2.236 (13.0128) | 1.659 (2.4584)
  25 minutes post dose 2 (n=48,47,36) | 0 (0.8858) | 1.845 (2.8085) | 3.325 (2.3515)
  2 hours post dose 1 (n=50,51,38) | 0 (0.0000) | 1.885 (1.7035) | 4.189 (2.8207)
  6 hours post dose 1 (n=50,50,37) | 0 (0.8899) | 0.874 (1.1988) | 2.818 (1.7195)

ADVERSE EVENTS:
Groups:
- Levalbuterol 0.63 mg: The experience of participants when treated with levalbuterol during the cross-over portion of the study.
- Arformoterol 7.5 Mcg: The experience of participants when treated with arformoterol 7.5 mcg during the cross-over portion of the study.
- Arformoterol 15 Mcg: The experience of participants when treated with arformoterol 15 mcg during the open-label portion of the study.
Arm/Group | Levalbuterol 0.63 mg | Arformoterol 7.5 Mcg | Arformoterol 15 Mcg
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/40
Other Adverse Events (participants affected / at risk) | 10/51 | 7/52 | 8/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levalbuterol 0.63 mg (N=51) | Arformoterol 7.5 Mcg (N=52) | Arformoterol 15 Mcg (N=40)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Potassium Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size was determined outside of statistical considerations. All data recorded at/after Visit 8 for 6 subjects, misdosed with ARF 7.5mcg instead of ARF 15mcg in open-label period, were excluded from the planned efficacy, PK and safety analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.